CLINICAL TRIAL: NCT03141632
Title: Effects of GLP-1 Analogues on Fluid Intake in Healthy Volunteers - "The GATE-Study"
Brief Title: Effects of Glucagon Like Peptide 1 (GLP-1) Analogues on Fluid Intake
Acronym: GATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GATE
Record Dates: First submitted 2017-04-27; First posted 2017-05-05 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Thirst; Water-Electrolyte Imbalance
MeSH Terms: conditions — Water-Electrolyte Imbalance | interventions — dulaglutide; calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo control, cross-over design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dulaglutide (Active Comparator): Dulaglutide (Trulicity®) 1.5 mg in 0.5 ml, via Pen s.c. once weekly for 3 weeks.
  Interventions: Drug: Dulaglutide
- Placebo (Placebo Comparator): 0.5 ml normal saline (0.9% sodium chloride), sc once weekly for 3 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dulaglutide — Evaluation visit with assessment of fluid intake
  Other Names: Verum
  Arms: Dulaglutide
Other: Placebo — Evaluation visit with assessment of fluid intake
  Arms: Placebo

SUMMARY:
The aim of this study is to elucidate whether GLP-1 analogues influence not only appetite but also thirst perception. It is hypothesized that GLP-1 analogues reduce fluid intake in healthy volunteers compared to Placebo.

DETAILED DESCRIPTION:
GLP-1 analogues are well known to stimulate glucose-induced insulin secretion and to reduce energy intake. Recent findings from animal and human studies suggest a role of GLP-1 in regulating water and salt homeostasis. GLP-1 has been shown to reduce fluid intake after an oral salt load or during a meal - pointing to a hypodipsic effect. The aim of this study is to elucidate whether these putative hypodipsic properties of GLP-1 analogues reduce fluid intake in healthy volunteers compared to placebo assessed during an evaluation visit of 8 hours.

ELIGIBILITY:
Inclusion Criteria:

- Age 18 to 65 years

Exclusion Criteria:

* Known or probable central or nephrogenic Diabetes insipidus, based on patient's history
* Polyuria secondary to diabetes mellitus, hypokalemia, hypercalcemia
* Primary Polydipsia, defined as more than 4 liters fluid intake per day
* BMI <18 or >30kg/m2
* Pregnancy
* Previous treatment with GLP-1 agonists within the last 3 month
* History of pancreatitis
* Severe renal insufficiency (eGFR (CKD EPI) <30 ml/min/1,73 m2)
* Cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05-12 (Actual)

PRIMARY OUTCOMES:
Fluid intake | 8 hours
  Fluid intake (ml) during an evaluation visit

SECONDARY OUTCOMES:
Thirst | 8 hours
  Thirst perception
Urine volume | 24 hours
  Urine volume in ml
Urinary sodium | 24 hours
  Urinary sodium excretion
Electrolytes | 3 timpoints during 8 hours
  Plasma electrolytes
Urine electrolytes | 3 timpoints during 8 hours
  Urine electrolytes
copeptin | 3 timpoints during 8 hours
  copeptin values
renin | 3 timpoints during 8 hours
  renin
aldosterone | 3 timpoints during 8 hours
  aldosterone
Water and Salt | 3 timpoints during 8 hours
  Brain Natriuretic Peptide (BNP)
GLP-1 | 3 timpoints during 8 hours
  GLP-1
Hypothalamus Pituitary Adrenal Axis (HPA) | 8 hours after Dexamethasone intake
  cortisol value after Dexamethasone intake
circadian rhythm | 16 hours
  circadian rhythm of serum cortisol
salivary cortisol | 16 hours
  circadian rhythm of salivary cortisol
ACTH | 16 hours
  circadian rhythm of ACTH
Hypothalamus Pituitary Adrenal Axis (HPA) | 0.5 hours
  cortisol upon adrenocorticotropic hormone (ACTH) stimulation
Hypothalamus Pituitary Adrenal Axis (HPA) | 24 hours
  free urinary cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof, Principal Investigator — University Hospital fo Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vukajlovic T, Sailer CO, Asmar A, Jensen BL, Vogt DR, Christ-Crain M, Winzeler B. Effect of a 3-Week Treatment with GLP-1 Receptor Agonists on Vasoactive Hormones in Euvolemic Participants. J Clin Endocrinol Metab. 2022 May 17;107(6):e2581-e2589. doi: 10.1210/clinem/dgac063. PMID 35134170